CLINICAL TRIAL: NCT01626924
Title: A Multi-centre, Randomised, Double-blind, Placebo-controlled Phase II Study to Evaluate the Efficacy, Safety, Tolerability and Pharmacokinetics of 2-Iminobiotin (2-IB) in Neonates With ≥36 Weeks GA With Moderate to Severe Perinatal Asphyxia
Brief Title: A Study of 2-Iminobiotin in Neonates With Perinatal Asphyxia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment too slow and site decided to use hypothermia (exclusion criteria)
Sponsor: Neurophyxia B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU 01-02-01; 2011-002502-74 (EudraCT Number)
Record Dates: First submitted 2012-06-15; First posted 2012-06-25 (Estimated); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Perinatal Asphyxia
Keywords: Perinatal Asphyxia; Neonatal encephalopathy; Oxygen shortage at birth; Antenatal asphyxia; hypoxia-ischaemia; birth asphyxia; asphyxia neonatorum
MeSH Terms: conditions — Asphyxia Neonatorum | interventions — 2-iminobiotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2-Iminobiotin (Experimental)
  Interventions: Drug: 2-Iminobiotin

INTERVENTIONS:
Drug: 2-Iminobiotin — 2-Iminobiotin is formulated as a 0.75 mg/ml isotonic, iso-osmotic, saline solution with a pH of 4. It is administered as a solution for I.V.infusion through a central catheter. Six pulse doses will be given in 20 hours. Dosage will starts with 0.2 mg/kg/dose, but may be adapted during the study.

SUMMARY:
In case of insufficient oxygen supply to the brain of a newborn child (perinatal asphyxia), toxic compounds will be formed. These toxic compounds will damage the cells of the brain. 2 Iminobiotin (2 IB) is an investigational medicinal product that is related to vitamin B7. From studies in animals it has been shown that 2-IB may prevent the formation of the toxic compounds. Also it has been shown to be safe in in studies in juvenile animals and in healthy, adult male volunteers. The doctors hope that this will prevent (part of) the potential brain damage that may result from lack of oxygen to the brain.

This study is the first study in the target population: newborn with moderate to severe oxygen shortage during birth. In this study the investigators evaluate short term efficacy, safety and pharmacokinetics of 2-Iminobiotin. In the follow-up phase the investigators evaluate the long term efficacy and safety.

The study hypothesis is that 2-Iminobiotin will help to decrease the brain damage after oxygen shortage and is indeed safe. The brain damage will be measured both in the first week and during the first two years of life. The study was designed as a study with two parts an open label pilot part (6 patients) and a double-blind randomised part (60 patients). Due to lack of recruitment it was decided in September2014 to stop recruitment after the open label pilot part of the study (6 patients).

ELIGIBILITY:
Inclusion Criteria:

1. Neonates with ≥ 36 and <44 weeks gestation with at least one of the following:

   * Apgar Score ≤ 5 at 10 minutes after birth
   * Continued need for resuscitation, including endotracheal or mask ventilation at 10 minutes after birth
   * Acidosis, defined as either umbilical cord pH or any arterial, venous, capillary pH within 60 minutes of birth pH ≤ 7.00
   * Acidosis, defined as base deficit ≥ 16 mmol/l in umbilical blood sample or any blood sample within 60 minutes of birth (arterial or venous).
2. The presence of moderate/severe encephalopathy defined as:

   * Altered state of consciousness (lethargy, stupor, coma) and at least one of the following:

     * Hypotonia
     * Abnormal reflexes including oculomotor or papillary abnormalities
     * Weak or absent suck reflex
     * Clinical seizures AND
   * Depression of the background pattern (lower margin≤ 5 µV meaning at least DNV or BS, CLV, FT) or the presence of seizure activity on the aEEG, registered for at least 30 minutes within 6h after birth.
3. Presence in hospital and ability to start treatment within 6h after birth.
4. Informed Consent Form signed before first study-related activity according to local law.
5. Receiving standard therapy without hypothermia.

Exclusion Criteria:

1. Major antenatally known- or congenital abnormalities, such as hernia diaphragmatica requiring ventilation.
2. Major antenatally known chromosomal abnormalities, such as trisomy 13 or 18 or neonates with evident syndromal appearances including brain dysgenesis.
3. Severe growth restriction with a birth weight below the 3rd percentile.
4. Inability to insert an indwelling catheter (umbilical venous catheter or percutaneously inserted central catheter, preferably multiple lumen).

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2012-06; Primary Completion 2014-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The Lac/NAA ratio in the basal ganglia as measured by single or multiple voxel Magnetic Resonance Spectroscopy (MRS). | The MRS will be performed between 3-7 days after birth
  Proton (1H) MRS of the basal ganglia lactate/N-acetyl aspartate (Lac/NAA) peak-area ratio is considered to be an accurate quantitative biomarker for prediction of neurodevelopmental outcome after Neonatal Encephalopathy (Thayyil et al, 2010). Results will be compared between arms.
The composite endpoint of survival at 48h with a normal aEEG | 48h after start treatment
  Electrocortical brain activity is measured by aEEG, starting as soon as possible after birth and before study medication has been initiated and continued until at least 72h after start of treatment. Every 4h the background pattern of the aEEG and the presence of seizures will be recorded in the eCRF. The aEEG will be classified as normal or abnormal at 48h after the start of treatment. Hence, for this primary endpoint, a good outcome is defined as survival in combination with a normal aEEG at 48h. A bad outcome is either death or abnormal aEEG at 48h after start treatment.

SECONDARY OUTCOMES:
MRI: pattern of injury score | The MRI will be performed between 3-7 days after birth
  Neuro-imaging by Magnetic Resonance Imaging (MRI) between 3 and 7 days following birth. The scoring system used is the pattern of injury score (Rutherford et al, 2010, appendix) in 4 areas of the brain (cortex, basal ganglia and thalamus, white matter and posterior limb of the internal capsule (PLIC)). Abnormal MRI is reported to be a predictor of poor outcome when at least one of following occurs (Rutherford et al, 2010):
  * Moderate or severe score in basal ganglia and thalamus
  * Abnormal PLIC
  * Severe white matter abnormalities Results will be compared between arms.
MRI: DWI (diffusion weighted images): apparent diffusion coefficient (ADC) in basal ganglia and PLIC | The MRI will be performed between 3-7 days after birth
aEEG. Background pattern | Every 4 hours until 48 hours after start treatment
  aEEG background will be evaluated every 4 hours until at least 48 hours after start treatment and also at time point of 48h after birth.
Mortality | first 7 days after birth
Length of stay at the level III NICU | On the average this is expected to be 4-14 days after birth
Neurodevelopmental status | 3,6,12,18 and 24 months after treatment
  During the follow-up visits the neurodevelopmental development is measured using age specific standardized tests, including AIMS, BSID-III, CBCL, general movements
Long term safety | 3,6,12,18,24 months
  During the follow-up period Serious Adverse Events are reported.
Safety during hospitalization period | Participants will be followed up for the duration of stay at hospital after birth (hospitalization period), on the average this will be 2-4 weeks
  During the hospitalization period a number of safety parameters are measured and compared between groups, including blood tests (blood gas, haematology, biochemistry), urinalysis, vital signs, fluid balance, clinical evaluation, local tolerance, growth parameters, EEG, ECG. Also number and kind of Adverse Events and Serious Adverse Events will be compared between arms.
Pharmacokinetics during the treatment phase | From start of treatment untill right after last treatment has been given (20h15min after start treatment)
  Pharmacokinetic parameters to be evaluated include:
  * Cmax (observed maximum plasma concentration)
  * AUC0-4h (area under the plasma concentration-time curve from time 0 to 4h after administration)
  * AUC0-∞ (area under the plasma concentration-time curve from time 0 to infinity)
  * T(end of infusion) (time at maximum plasma concentration).
  * t1/2 (terminal elimination half-life)
  * CL (clearance)
  * V (volume of distribution)
Neurological status as assessed by full neurological examination | at discharge from level III NICU on the average this will 7-14 days after birth.
  Full neurological examination includes:
  Prechtl state, Higher cortical functions, Pupillary reflexes right,Pupillary reflexes left, corneal reflex right, corneal reflex left, optokinetic reflexes, nystagmus, facial symmetry, tone, spontaneous movements right, spontaneous movements left, tendon reflexes, ankle clonus right, ankle clonus left, sucking reflex, grasp reflex right, grasp reflex left, moro reflex right, moro reflex left, glabella reflex, snout reflex, palmomental reflex right, palmomental reflex left. Outcomes will be compared between arms
aEEG. Time to normal aEEG | Up to 72 hours after start treatment
  The time to normal aEEG will be determined for each subject.
aEEG. Seizures (clinical and sub-clinical) | 48 hours after start treatment
  The number and severity of clinical and sub-clinical seizures will be evaluated for each subject.
aEEG. Time to normal sleep-wake cycling | up to 72 hours after start treatment
  The time to normal sleep-wake cycling will be determined for each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Leufkens, PharmD, Study Director — Neurophyxia B.V.
Locations (2):
- Turkey (Türkiye) (2):
  - T.R. Ministry of Health Izmir Tepecik Training and Research Hospital, Izmir
  - Yıl University Medical Faculty Hospital, Van

REFERENCES:
- [Background] Peeters-Scholte C, Koster J, Veldhuis W, van den Tweel E, Zhu C, Kops N, Blomgren K, Bar D, van Buul-Offers S, Hagberg H, Nicolay K, van Bel F, Groenendaal F. Neuroprotection by selective nitric oxide synthase inhibition at 24 hours after perinatal hypoxia-ischemia. Stroke. 2002 Sep;33(9):2304-10. doi: 10.1161/01.str.0000028343.25901.09. PMID 12215603